CLINICAL TRIAL: NCT02835755
Title: Increasing HPV Vaccine Coverage Among Young Adult Gay and Bisexual Men
Brief Title: Mobile Health Intervention in Increasing HPV Vaccine Coverage Among Young Adult Gay and Bisexual Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Reiter, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-15234; NCI-2016-00819 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH); R21CA194831 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-18 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Control) (Active Comparator): Patients receive standard information about HPV and HPV vaccine, such as the VIS, on a mobile-friendly website study portal.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Group II (mHealth HPV vaccine) (Experimental): Patients receive the mHealth HPV vaccine intervention consisting of content about HPV and HPV vaccine on the study portal for 15 minutes and vaccination reminders sent by the portal via text or e-mail.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive standard HPV and HPV vaccine information
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (Control)
Other: Educational Intervention — Receive mHealth HPV vaccine intervention
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (mHealth HPV vaccine)
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot trial studies how well a mobile health (mHealth) human papillomavirus (HPV) vaccine intervention works in increasing HPV vaccine coverage among young adult gay and bisexual men. Giving young men information about the HPV vaccine and the importance of vaccination may encourage them to get the HPV vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Pilot test a mobile health (mHealth) HPV vaccine intervention for young gay and bisexual men to establish feasibility and acceptability.

II. Obtain preliminary efficacy data on whether the mHealth HPV vaccine intervention increases HPV vaccine initiation compared to the control group.

SECONDARY OBJECTIVES:

I. Examine whether the mHealth HPV vaccine intervention affects secondary outcomes compared to the control group.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (CONTROL): Patients receive standard information about HPV and HPV vaccine, such as the vaccine information statement (VIS), on a mobile-friendly website study portal.

GROUP II (INTERVENTION): Patients receive the mHealth HPV vaccine intervention consisting of content about HPV and HPV vaccine on the study portal for 15 minutes and vaccination reminders sent by the portal via text or e-mail.

All patients complete a survey on the study portal at baseline, immediately after the mHealth intervention or control materials, and at 3 months and 7 months thereafter for about 10-15 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as gay or bisexual
* Lives in the United States (US)
* Has not received any doses of HPV vaccine

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2017-04-16 (Actual)

PRIMARY OUTCOMES:
Acceptability will be established by examining participant satisfaction with study materials | Up to 7 months
  Linear regression will be used and usage data and satisfaction with vaccination reminders (intervention group only) will be descriptively examined.
Feasibility established by achieving recruitment, retention, and medical record release goals | Up to 7 months
  Critical parameters with point estimates and 95% confidence intervals will be estimated and tested with a two-sided alpha=.05
Receipt of 1 or more doses of HPV vaccine | Up to 7 months
  Evaluated using logistic regression.

SECONDARY OUTCOMES:
Changes in potential mediators between study group and HPV vaccination (i.e., protection motivation theory [PMT] constructs and HPV and HPV vaccine knowledge) | Up to 7 months
  Evaluated using analysis of covariance models.
Receipt of second and third doses of HPV vaccine | Up to 7 months
  Evaluated using logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Reiter, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Reiter PL, Katz ML, Bauermeister JA, Shoben AB, Paskett ED, McRee AL. Increasing Human Papillomavirus Vaccination Among Young Gay and Bisexual Men: A Randomized Pilot Trial of the Outsmart HPV Intervention. LGBT Health. 2018 Jul;5(5):325-329. doi: 10.1089/lgbt.2018.0059. PMID 29979642
- [Derived] McRee AL, Shoben A, Bauermeister JA, Katz ML, Paskett ED, Reiter PL. Outsmart HPV: Acceptability and short-term effects of a web-based HPV vaccination intervention for young adult gay and bisexual men. Vaccine. 2018 Dec 18;36(52):8158-8164. doi: 10.1016/j.vaccine.2018.01.009. Epub 2018 Jan 10. PMID 29331245
- See also: The Jamesline — http://cancer.osu.edu